CLINICAL TRIAL: NCT02499484
Title: The Use of Topical Glyceryl Trinitrate (GTN) and Eccentric Exercises in the Treatment of Midportion Achilles Tendinopathy: a Randomized Placebo Controlled Trial
Brief Title: Topical Glyceryl Trinitrate (GTN) and Eccentric Exercises in the Treatment of Midportion Achilles Tendinopathy
Acronym: NEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCSI-1764
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2018-04

CONDITIONS: Tendinopathy; Achilles Tendon Pain
MeSH Terms: conditions — Tendinopathy | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GTN and eccentric exercises (Active Comparator): Participants will complete a 12 week eccentric exercise program and use 0.5cm of glyceryl trinitrate ointment daily for 24 weeks
  Interventions: Drug: glyceryl trinitrate; Other: Eccentric exercise program
- Placebo and eccentric exercises (Placebo Comparator): Participants will use a placebo ointment with no active ingredient for 24 weeks and complete an eccentric exercise program for 12 weeks
  Interventions: Other: Placebo ointment; Other: Eccentric exercise program

INTERVENTIONS:
Drug: glyceryl trinitrate — Topical GTN will be used daily in combination with a eccentric home exercise program
  Other Names: Percutol
  Arms: GTN and eccentric exercises
Other: Placebo ointment — Topical placebo ointment will be used in combination with a eccentric home exercise program
  Other Names: aqueous cream
  Arms: Placebo and eccentric exercises
Other: Eccentric exercise program — All participants will complete the eccentric exercise program as a home exercise program daily.
  Other Names: Alfredson's eccentric exercise program

SUMMARY:
The primary objective of this research is to determine if the addition of topical GTN over 24 weeks to a 12 week exercise programme improves clinical outcomes more than placebo GTN for people with Achilles Tendinopathy.

Pain in the Achilles tendon is a common condition seen by physiotherapists and doctors. It affects people involved in sports and those who are not. It can limit the ability to walk, hop, jump and run. If the pain persists for longer than 3 months it can become extremely difficult to abolish. As a result, people with this common condition can suffer from prolonged pain and often the pain will persist and affect everyday activities.

While this is an easy injury to diagnose, it is not so easy to treat. Many treatments do exist, but often just provide short-term relief until the pain returns. Specific strengthening exercises have been shown to be beneficial in treating this condition.

The current project will study Achilles tendon pain in Irish adults at Connolly Hospital, Dublin, and will take place from 2015 to 2019. In this study, there are two groups of patients. Both groups will perform an exercise program for 12 weeks. Physiotherapists will instruct them on how to perform the exercises. Each group will be given an ointment to place on the sore tendon using an applirule. This ointment will be applied daily for 6 months. One group will use an ointment containing nitroglycerin, the other group will use an ointment with no active ingredient. This is called a placebo. The patients will apply the ointment daily for 6 months.

The patients will be assessed at the start of the program and after 6, 12 and 24 weeks. Our main question is to see whether this exercise program when combined with a nitroglycerin ointment applied directly over the sore tendon can improve the outcomes and recovery time for people who suffer with Achilles tendon pain.

DETAILED DESCRIPTION:
Study Design

The study will be designed to meet CONSORT guidelines. A randomized placebo controlled trial will be carried out at the Physiotherapy Department of Connolly Hospital, Blanchardstown, Dublin 15. The study will be conducted on patients who present to the department with a diagnosis of Achilles tendinopathy. The diagnosis will be confirmed based on a history of an insidious onset of Achilles tendon pain, a tender nodule/thickening of the tendon to the region 2 to 6cm from the calcaneal insertion, and an ultrasound examination that excludes a frank tear.

Participants will be randomly allocated to one of 2 groups. Group 1 will receive GTN for 24 weeks in combination with a supervised eccentric exercise programme delivered over 12 weeks. Group 2 will receive placebo GTN in addition to the same exercise programme.

Ethical Considerations Ethics approval will be sought from Connolly Hospital Research and Ethics Committee. All participants will give written informed consent.

At the patient's initial assessment, the following will be completed

* Outcome measure questionnaires - Victorian Institute of Sport Assessment-Achilles (VISA-A), Lower Extremity Functional Scale (LEFS), Numeric Rating Scale for pain (NRS)
* Assessment of Achilles tendon tenderness using pressure algometry
* Ultra-sound assessment of the Achilles tendon - tendon thickness measurements
* Proprioception testing (modified Star Excursion Balance Test)
* Simple strength tests of the Achilles, Hopping and heel raises

It is anticipated that the baseline assessment will take 60-75 minutes to complete. The follow-up assessment should take no more than 45 minutes to complete.

Outcome Measures All outcomes will be administered at baseline, and at week 6, 12 and 24 by the principal investigator. Data on adverse effects, compliance with the ointment application and the exercise program will be recorded at these scheduled visits.

Upon completion of the initial assessment by the principal investigator, participants will be scheduled to have their first exercise intervention session with one of the physiotherapists in Connolly Hospital. The treating physiotherapists will be trained in the exercise protocol and will be blinded to the type of GTN provided to the patient. This appointment will be scheduled within one week of the lead investigator's assessment. This tendon rehabilitation program is designed to encompass current methods of non-operative treatment of Achilles tendinopathy (Paoloni et al, 2004) and will involve the following:

* Instruction in performance of the Alfredson heavy load eccentric exercise program.
* Patients will be advised to avoid weight bearing sporting activities for the first 4 to 6 weeks, after which time gradual return to sports will be encouraged. Participation in sports will be continued so long as the pain does not increase above NRS>3 and no increase in Achilles morning stiffness is experienced.
* Instruction in the performance of daily static stretches of the gastrocnemius and soleus muscle groups
* Patients will be advised to avoid the use of co-interventions or complimentary treatments for the duration of the study.

Exercise interventions:

Participants will be instructed on how to perform the Alfredson heavy load eccentric exercise protocol (Alfredson, 1998) by the physiotherapists in Connolly Hospital. This will be performed during their first treatment session, which will take place approximately one week after the initial assessment. The participants will be given practical instructions and a written manual on the exercise program, which will include advice on progression of the exercise regimen.

Topical nitroglycerin ointment (GTN)

The topical GTN to be used for the purpose of this trial is Percutol. This will deliver the GTN in ointment form. Participants will be instructed in how to measure 0.5cm of Percutol ointment by applying 0.5cm of Percutol to a paper applicator/strip, which has the amount required indicated in a circular outline, measuring approximately the same size as a pea. This paper applicator/strip will be placed on a flat surface and the participant will squeeze the ointment onto the paper, carefully measuring the amount specified on the paper applicator. Participants will then place the paper on to the painful area of the Achilles with the ointment contacting the skin, and use the paper to lightly spread the ointment to cover the painful area of the Achilles tendon. The ointment should not be rubbed into the skin. The paper applicator will then be covered with surgical tape to hold the applicator in place. The participants will then replace the cap on the ointment and screw it on tightly and store it as per the instructions (at room temperature and out of reach and sight of children). Participants will be instructed to wash their hands before and after this process. The paper applicator with the Percutol ointment will be placed on the affected area of the Achilles tendon in the morning and left in situ for the daytime, and removed by the participant before sleeping at night. It will be emphasized that the ointment must be on while the participants perform the home exercise program (HEP).

0.5cm of Percutol has been chosen for the purpose of this trial. Aspire Pharma United Kingdom (UK) manufacture Percutol and have informed the PI that 1 inch of Percutol weighs 0.83g approximately and corresponds to 16.64mg of GTN.

The PI has conducted measures of Percutol, 0.5cm of Percutol weighs approximately 0.14 to 0.17g and this corresponds to 2.8 to 3.4mg of GTN.

The placebo to be used for the purpose of this trial will be aqueous cream and therefore will contain no GTN or active ingredient, which would assist in tendon healing. Participants will be instructed to apply the same amount of this placebo ointment in the exact same method as outlined for the GTN group using the same paper/applicator method.

Participants will be instructed in the use of the ointment during their initial visit with the lead investigator. They will be informed that the dosing regimen calls for the ointment to be applied to the painful area of the Achilles tendon and left in situ for 12 to 14 hours and removed at night prior to sleeping. This will then be discarded and replaced with a new measure of the ointment the next day. Participants will be advised to apply the ointment to the site of maximal tenderness within a region of 1-2 cm around this point. The participants will be advised to rotate the paper applicator about the site of maximal tenderness on a regular basis for the six-month duration of the study in an effort to minimize irritation of the skin.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of Achilles tendinopathy
2. Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol
3. Subjects must be male or female, aged 18 years or above at Baseline
4. Achilles pain of >3 months or more
5. Mid-portion Achilles tenderness and thickening on palpation
6. Confirmation of the diagnosis upon Ultra-sound assessment, and ruling out of other pathologies (eg: ruptures)

Exclusion Criteria:

1. Previous corticosteroid injection to the affected tendon in the past 3 months
2. Symptoms of less than 3 months duration
3. Previous use of topical GTN
4. Current use of nitrates, eg: GTN spray, tablet, transdermal patch.
5. Contra-indication to GTN therapy (see section 12.2.3)
6. Current pregnancy, breastfeeding or planning pregnancy
7. VISA-A score > 80
8. Previous surgery to the affected Achilles tendon
9. Seronegative spondyloarthropathy with Achilles enthesitis
10. Previous performance of a heavy load eccentric exercise program of the Achilles in the last 2 years
11. Severe migraines which fail to respond to over the counter medication and require specific migraine management
12. Inability to perform the exercise program due to serious illness, such as unstable angina/blood pressure, myocardial infarction in past three months, cardiomyopathy, uncontrolled metabolic disease, recent ECG changes, advanced respiratory disease or third degree heart block.
13. Any medical or psychiatric condition that the investigator deems appropriate for exclusion
14. Staff or students of Connolly Hospital, Blanchardstown

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-09; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
VISA A, Victoria Institute of Sport Assessment - Achilles | Change from baseline in VISA A at week 6,12 and 24
  The primary outcome will be the Victoria Institute of Sport Assessment, Achilles (VISA-A) scale, which measures the impact of Achilles tendinopathy on individuals' lifestyle. The VISA-A is a valid, reliable and user friendly self-report index of severity of Achilles tendinopathy (score 0 = worst, score 100 =perfect), can be easily administered in clinical practice (Robinson et al, 2001) and has been used as an outcome measure in other tendinopathy trials (Tumilty et al, 2012).

SECONDARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) | Baseline and week 6, 12 and 24
  The LEFS is a self-report measure of functional ability in relation to their Achilles tendinopathy, which will be completed by participants. The LEFS has been shown to have good construct validity and reliability. It is easy to administer and score so is applicable for research purposes and clinical decision making for individual patients (Binkley et al., 1999).
Pain Detection Threshold, PDT using pressure algometry | baseline and week 6, 12 and 24
  The outcome measurement in pressure algometry is the pain detection threshold (PDT), measured in kg/f, or the point at which pressure pain is first experienced by the participant. As tenderness is one of the key clinical diagnostic criteria, algometry is an appropriate measure to quantify the pain pressure response.
Ultra sound measure of Achilles thickness | Baseline and week 6, 12 and 24
  Ultra sound will be used to measure any change in transverse thickness (measure in mm) of the achilles over the course of the trial
Numeric Rating Scale (NRS) for pain | Baseline and week 6, 12 and 24
  Participants will be asked to rate their Achilles pain from zero to ten on a numerical rating scale (NRS). Standardized and validated pain scales provide a means of measuring a patient's pain and of evaluating the response to treatment. Williamson and Hogart (2005) determined that NRS is valid, reliable and appropriate for use in clinical practice. Participants will be asked to verbally rate their level of perceived pain intensity on a numerical scale from 0 to 10, with zero representing "no pain" and 10 representing the "the worst pain possible"
Star Excursion Balance Test (SEBT) | baseline and week 6, 12 and 24
  The modified Star Excursion Balance Test (SEBT) will be performed to assess whether any difference exists between the 2 groups and between the affected and unaffected limbs. The SEBT (appendix 3) has been shown to be a reliable measure of dynamic balance (Hertel et al, 2006).
Heel raise for endurance | Change in number of heel raises performed at baseline and week 6, 12 and 24
  The heel raise test for endurance will be performed on one leg at a time with the participant standing. The participant will be allowed to have two fingers per hand, placed at shoulder height, against a wall for balance. Participants will be instructed to raise up as high as possible onto the toes and then lower the heel to the starting position and repeat this technique for as many as possible on each leg. The test will be terminated when the patient stops, or can no longer perform a heel raise. The number of heel raises and any pain associated with the test will be documented using the NRS.
Heel raise for endurance | Change in NRS with heel raises performed at baseline and week 6, 12 and 24
  The heel raise test for endurance will be performed on one leg at a time with the participant standing. The participant will be allowed to have two fingers per hand, placed at shoulder height, against a wall for balance. Participants will be instructed to raise up as high as possible onto the toes and then lower the heel to the starting position and repeat this technique for as many as possible on each leg. The test will be terminated when the patient stops, or can no longer perform a heel raise. The number of heel raises and any pain associated with the test will be documented using the NRS.
Hopping tests | Change in number of hops performed at baseline and weeks 6, 12 and 24
  Hopping tests involve the stretch shortening cycle of the Achilles tendon and calf musculature, and therefore measure the muscle tendon units elastic properties. Participants will be instructed to perform hopping on one leg at a time, with arms by the side, in a natural rhythm. A natural jump frequency is approximately 2 hops per second. Participants will be instructed to perform 20 hops on each leg with 15 to 30 seconds rest between each side. The number of hops performed and pain associated with hopping on each side will be documented using the NRS.Both the heel raise to endurance and hopping test have been shown to reliable tests with good test-retest reliability in previous studies of Achilles tendinopathy (Silbernagel et al, 2001 and 2006).
Hopping tests | Change in NRS associated with hopping performed at baseline and weeks 6, 12 and 24
  Hopping tests involve the stretch shortening cycle of the Achilles tendon and calf musculature, and therefore measure the muscle tendon units elastic properties. Participants will be instructed to perform hopping on one leg at a time, with arms by the side, in a natural rhythm. A natural jump frequency is approximately 2 hops per second. Participants will be instructed to perform 20 hops on each leg with 15 to 30 seconds rest between each side. The number of hops performed and pain associated with hopping on each side will be documented using the NRS. Both the heel raise to endurance and hopping test have been shown to reliable tests with good test-retest reliability in previous studies of Achilles tendinopathy (Silbernagel et al, 2001 and 2006).

CONTACTS AND LOCATIONS:
Overall Officials: Helen French, PhD, Study Director — Royal College of Surgeons, Ireland; Trevor Duffy, MD, MBA, Study Director — Connolly Hospital, Dublin 15, Ireland
Locations (1):
- Connolly Hospital, Blanchardstown, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paoloni JA, Appleyard RC, Nelson J, Murrell GA. Topical glyceryl trinitrate treatment of chronic noninsertional achilles tendinopathy. A randomized, double-blind, placebo-controlled trial. J Bone Joint Surg Am. 2004 May;86(5):916-22. doi: 10.2106/00004623-200405000-00005. PMID 15118032
- [Background] Alfredson H, Pietila T, Jonsson P, Lorentzon R. Heavy-load eccentric calf muscle training for the treatment of chronic Achilles tendinosis. Am J Sports Med. 1998 May-Jun;26(3):360-6. doi: 10.1177/03635465980260030301. PMID 9617396
- [Background] Robinson JM, Cook JL, Purdam C, Visentini PJ, Ross J, Maffulli N, Taunton JE, Khan KM; Victorian Institute Of Sport Tendon Study Group. The VISA-A questionnaire: a valid and reliable index of the clinical severity of Achilles tendinopathy. Br J Sports Med. 2001 Oct;35(5):335-41. doi: 10.1136/bjsm.35.5.335. PMID 11579069
- [Background] Tumilty S, McDonough S, Hurley DA, Baxter GD. Clinical effectiveness of low-level laser therapy as an adjunct to eccentric exercise for the treatment of Achilles' tendinopathy: a randomized controlled trial. Arch Phys Med Rehabil. 2012 May;93(5):733-9. doi: 10.1016/j.apmr.2011.08.049. PMID 22541305
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Hertel J, Braham RA, Hale SA, Olmsted-Kramer LC. Simplifying the star excursion balance test: analyses of subjects with and without chronic ankle instability. J Orthop Sports Phys Ther. 2006 Mar;36(3):131-7. doi: 10.2519/jospt.2006.36.3.131. PMID 16596889
- [Background] Silbernagel KG, Gustavsson A, Thomee R, Karlsson J. Evaluation of lower leg function in patients with Achilles tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2006 Nov;14(11):1207-17. doi: 10.1007/s00167-006-0150-6. Epub 2006 Jul 21. PMID 16858560
- [Background] Silbernagel KG, Thomee R, Thomee P, Karlsson J. Eccentric overload training for patients with chronic Achilles tendon pain--a randomised controlled study with reliability testing of the evaluation methods. Scand J Med Sci Sports. 2001 Aug;11(4):197-206. doi: 10.1034/j.1600-0838.2001.110402.x. PMID 11476424
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093